CLINICAL TRIAL: NCT00684710
Title: Ascending Single Dose Study of the Safety, Tolerability, and Pharmacokinetics of PAZ 417 Administered Orally to Healthy Young Japanese Male and Healthy Elderly Japanese Male Subjects
Brief Title: Study Evaluating the Safety, Tolerability and Activity of One Dose of PAZ-417 Given to Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3186A1-101
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Alzheimer Disease; Healthy
Keywords: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PAZ-417 (Experimental)
  Interventions: Drug: PAZ-417
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PAZ-417
  Arms: PAZ-417
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will provide an initial assessment of the safety, tolerability, and pharmacokinetics (PK) of PAZ-417 after administration of ascending single oral doses to healthy young Japanese male and healthy elderly Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria

1. Men aged 20 to 45 years inclusive (healthy young male subjects) and ≥65 years inclusive (healthy elderly male subjects)
2. Nonsmoker or smoker of fewer than 10 cigarettes per day.
3. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG).

Exclusion Criteria

1. Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
2. Subjects who are identified as being at risk for hypercoagulability
3. Use of any investigational or prescription drug within 30 days before test article administration

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 3 months

SECONDARY OUTCOMES:
Pharmacokinetics | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Kitashinagawa, Shinagawa-ku, Tokyo, Japan